CLINICAL TRIAL: NCT06214624
Title: Effects of Exercise on Brain Health in Patients With Coronary Heart Disease: the Heart-Brain Randomized Controlled Trial
Brief Title: Exercise and Brain in Coronary Heart Disease
Acronym: Heart-Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Instituto Mixto Universitario Deporte y Salud (iMUDS) (Unknown); Centro de Investigación Mente, Cerebro y Comportamiento (CIMCYC) (Unknown); University Hospital Virgen de las Nieves (Other); Hospital Clinico Universitario San Cecilio (Other); Centro de Investigación Biomédica en Red de la Fisiopatología de la Obesidad y Nutrición (CIBEROBN) (Unknown)
Responsible Party: Principal Investigator, Francisco B. Ortega Porcel, Full Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1776-N21
Record Dates: First submitted 2023-12-22; First posted 2024-01-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Heart Disease
Keywords: coronary artery disease; ischemic heart disease; exercise; HIIT; resistance training; brain; cognition; magnetic resonance imaging
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Myocardial Ischemia; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12-week of aerobic high-intensity interval training (HIIT) exercise program (Experimental)
  Interventions: Behavioral: Two types of exercise interventions
- 12-week aerobic HIIT plus resistance exercise program (Experimental)
  Interventions: Behavioral: Two types of exercise interventions
- Usual care, Wait-list control group (No Intervention): The control group (as well as the 2 intervention groups) will be treated as usual in outpatient Phase III, which in Spain includes periodic medical revisions and medication control. In addition, for the control group, we will apply the wait-list strategy providing the supervised exercise program once all data collection for pre- and post-intervention assessment points have been finished.

INTERVENTIONS:
Behavioral: Two types of exercise interventions — * HIIT. 3 times/week. This consists of a 4x4 HIIT (preferably in treadmill), 4 intervals of 4min at high intensity (85-95% HRmax) and 3 intervals of 3min of active resting at ~70% HRmax in between. All sessions including 10 min of warming-up and 10min of cooling down, resulting in 45min sessions. The first 2 weeks will progress from moderate-intensity training to HIIT for a better adaptation and acceptability of the program.
  * HIIT + resistance. 3 times/week. The aerobic part consists of a 3x4 HIIT (preferably in treadmill), 3 intervals of 4min at high intensity (85-95% HRmax) and 2 intervals of 3min of active resting (~70% HRmax) in between. The resistance part consists of 2 series of an 8-exercise circuit (combination of upper and lower body exercises using elastic bands and body weight) with a ratio of 20sec of effort - 40sec of resting. Sessions will have 5min of warming up in the treadmill and 5min of cooling down walking in the gym, comprising a total of 45min sessions.
  Arms: 12-week aerobic HIIT plus resistance exercise program; 12-week of aerobic high-intensity interval training (HIIT) exercise program

SUMMARY:
The Heart-Brain project is a randomized controlled trial designed to examine the effects of two different exercise programs of 12-week duration: 1) aerobic high intensity interval training (HIIT), and 2) aerobic HIIT plus resistance training, on brain health and other outcomes in coronary heart disease patients.

DETAILED DESCRIPTION:
Patients with coronary heart disease (CHD) has higher risk of developing dementia, cognitive impairment, and mental disorders. There is, therefore, a need to identify effective and sustainable initiatives to avoid or attenuate cognitive and mental health declines in these patients, and in this context, physical exercise can play a major role. The overall objective of the present project is to investigate the effects of exercise on brain health outcomes in CHD patients. The Heart-Brain project is a single-blinded, exercise-based randomized controlled trial. We will run a three-arms trial with a waiting-list control group, and two intervention groups that will receive two different supervised exercise programs: 1) aerobic high intensity interval training (HIIT) and 2) a combination of aerobic HIIT plus resistance training. The study will be conducted in 90 patients with CHD who meet the eligibility criteria indicated below.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 50 and 75 years old, both inclusive (*Contingency plan: increase the range to 40-75 if we have difficulties to get the study sample)
2. Must have stable coronary heart disease (phase III), proven by invasive coronary angiography or CT with at least one coronary lesion > 50%.
3. Able to speak and read fluent Spanish.
4. Live in Granada city or surrounding areas (able to come to evaluations and exercise program)
5. Living in community during the study (i.e. independent home, non-assisted living facilities)
6. Ejection fraction ≥ 45%.
7. Functional grade I-II according to the New York Heart Association (NYHA) scale.
8. Sinus rhythm.
9. Stable optimal medical treatment (3 or more drugs at the determined by a cardiologist).
10. Physically inactive, considering: 1) not meeting the WHO recommendations in both the aerobic and strength part, and 2) not to be participating in a planned and structured exercise program at least 3 days per week and for more than 3 months. Both conditions must be met to be included. Note: going for a walk will not be considered an exclusion reason.
11. Classified as cognitively normal according to Stics-m

Exclusion Criteria:

1. Used of assisted walking devices.
2. Acute coronary syndrome in the last year, coronary surgery, or percutaneous intervention in the last 6 months.
3. Treatment for any type of cancer in the last 2 years.
4. Severe hospitalization in the intensive care unit in the last 6 months.
5. Current psychiatric diagnosis (visit to psychiatrist and drug treatment prescription in the last year), including major depression and history of psychiatric illness (schizophrenia, bipolar disorder, hallucinations).
6. Grade III obesity.
7. Diagnosis of neurological or cerebrovascular disorder (e.g. stroke).
8. Medical contraindication for inclusion in an exercise program.
9. Diabetes with uncontrolled glycemia.
10. Resting blood pressure > 180/110.
11. Chest pain with exertion or changes in the ST segment suggestive of severe ischemia during ergometry.
12. Severe inducible ischemia
13. Functional capacity in ergometry (<5 METS).
14. Obstructive left main artery disease (significant disease > 50%)
15. Unstable angina
16. Uncontrolled cardiac arrhythmia
17. Presence of metal implants (e.g., pacemaker or implantable cardioverter-defibrillator-ICD) not compatible with MRI (reported during the phone screening)
18. Paroxysmal or persistent atrial fibrillation with episodes in the last 6 months.
19. Moderate to severe pulmonary hypertension.
20. Acute endocarditis, myocarditis, or pericarditis.
21. Moderate to severe valve disease (grade 3-4)
22. Acute pulmonary embolism, or deep vein thrombosis.
23. Aortic dissection
24. High-grade heart block or complete left bundle branch block or altered basal electrocardiogram with difficulties to interpret in exercise testing.
25. Hypertrophic obstructive cardiomyopathy.
26. Retinopathy.
27. Severe autonomic or peripheral neuropathy.
28. Acute systemic illness or fever.
29. Acute or chronic renal failure (estimated glomerular filtration rate < 30 mL/min)
30. Pulmonary fibrosis or interstitial disease (respiratory failure or severe COPD confirmed by pneumological study).
31. Recent treatment for alcohol or substance abuse.
32. Claustrophobia.
33. Any surgery or medical intervention planned during the study period.
34. Plans to participate or current participation in other studies that might interferes with this study.
35. Current pregnancy or intention to get pregnant during the study period

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow | Baseline and 12 weeks
  The main outcome is the change in global cerebral blood flow from baseline to 12 weeks. Cerebral blood flow will be measured using the magnetic resonance imaging technique of TGSE-pCASL (turbo gradient spin echo-pseudo continuous arterial spin labeling). Additionally, regional cerebral blood flow will be determined in a voxel-wise analysis to measure local perfusion.

SECONDARY OUTCOMES:
Change cerebral vascularization | Baseline and 12 weeks
  Cerebral vascularization will be measured using the magnetic resonance angiography TOF (Time-of-flight angiography).
Change in executive function and general cognition | Baseline and 12 weeks
  A comprehensive neuropsychological battery will assess several domains of executive function: working memory, cognitive flexibility and inhibitory control, and an executive function score will be computed and used as main behavioral outcome . Additionally, the general cognition will be assessed by the MOCA (MONTREAL COGNITIVE ASSESSMENT) test.
Change in cardiorespiratory fitness | Baseline and 12 weeks
  Cardiorespiratory fitness will be assessed by a cardiorespiratory exercise test in a treadmill measuring gas exchange (treadmill time-to-exhaustion and VO2peak)

OTHER OUTCOMES:
Change in blood brain barrier (BBB) permeability | Baseline and 12 weeks
  BBB permeability will be operationally measured by using a recently developed neuroimaging technique that measures water exchange across the BBB using 3D diffusion-prepared arterial spin labelled perfusion MRI.
Change in brain morphology | Baseline and 12 weeks
  MRI (magnetic resonance imaging) will measure brain morphology including volume, area, cortical thickness, and shapes by a T1-weighted MPRAGE structural sequence.
Change in white matter structure | Baseline and 12 weeks
  MRI (magnetic resonance imaging) will measure white matter structure and lesions by diffusion weighted acquisition sequence.
Change in brain function | Baseline and 12 weeks
  MRI (magnetic resonance imaging) will measure brain function during resting state. Measures of brain activity and brain connectivity will be calculated.
Change in blood-based neurology biomarkers | Baseline and 12 weeks
  Blood samples will be used to determine plasmatic concentration of peripheral neurology biomarkers including brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor (VEGF) and cathepsin B (CTSB), as well as novel neurodegenerative biomarkers based on new evidence up to the time of the analysis.
Change in saliva-based neurology biomarkers | Baseline and 12 weeks
  Saliva samples will be used to determine concentration of peripheral neurology biomarkers including brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor (VEGF) and cathepsin B (CTSB), as well as novel neurodegenerative biomarkers based on new evidence up to the time of the analysis.
Hemodynamic vascular changes | Baseline and 12 weeks
  Hemodynamic vascular parameters will be measured using ultrasound echography (i.e. carotid intima-media thickness).
Hemodynamic cardiac changes | Baseline and 12 weeks
  Cardiac parameters will be measured using ultrasound echography (i.e. ejection fraction, cardiac volumes, and cardiac output)
Hemodynamic transcranial changes | Baseline and 12 weeks
  Hemodynamic transcranial parameters will be measured using ultrasound echography (i.e. Doppler diastolic-systolic velocity).
Change in general muscular strength | Baseline and 12 weeks
  The maximum isometric strength of the hand and forearm muscles measured with the handgrip test (Kg) will be used to determine general muscular strength.
Change in lower body muscular strength | Baseline and 12 weeks
  Muscular strength in lower body will be assessed using the chair stand test (number of repetitions).
Change in upper body muscular strength | Baseline and 12 weeks
  Muscular strength in upper body will be assessed using the arm curl test (number of repetitions).
Change in physical function | Baseline and 12 weeks
  Senior Fitness Test (including the 6-min walking test) will assess overall physical functioning and z-scores will be calculated.
Change in depression | Baseline and 12 weeks
  Depressive symptoms will be assessed using the Global Deterioration Scale, the Health Survey Short Form (SF-36) and the Hospital Anxiety and Depression Scale.
Change in anxiety | Baseline and 12 weeks
  Anxiety will be assessed using the Health Survey Short Form (SF-36) and the Hospital Anxiety and Depression Scale.
Change in stress outcomes | Baseline and 12 weeks
  Stress outcomes will be assessed using the Perceived Stress Scale.
Change in loneliness | Baseline and 12 weeks
  Loneliness will be assessed using the UCLA Loneliness Scale.
Change in self-esteem outcomes | Baseline and 12 weeks
  Self-esteem will be assessed using the Rosenberg Self-Esteem Scale.
Change in social support outcomes | Baseline and 12 weeks
  Social support will be assessed using the Social Provisions Scale.
Change in health-related quality of life | Baseline and 12 weeks
  Global, physical, and mental health-related quality of life will be self-reported using the Health Survey Short Form (SF-36), in which higher scores means a better health-related quality of life.
Change in physical activity | Baseline and 12 weeks
  Physical activity will be measured using the accelerometer Axivity AX, and a self-reported questionnaire based on the Global Physical Activity Questionnaire.
Change in sedentary behaviors | Baseline and 12 weeks
  Sedentary behaviors will be measured using the accelerometer Axivity AX, and a self-reported questionnaire based on the Global Physical Activity Questionnaire.
Change in sleep quality | Baseline and 12 weeks
  Sleep quality will be measured using the accelerometer Axivity AX, and using the Pittsburgh Sleep Quality Index.
Change in diet behaviors | Baseline and 12 weeks
  Diet behaviors will be self-reported using the 14-item Questionnaire of Mediterranean Diet Adherence (PREDIMED-14), and a self-reported question for supplements intake.
Change in body mass index | Baseline and 12 weeks
  Body mass index (BMI) will be assessed using a dual-energy x-ray absorptiometer (DXA) and a TANITA's Bioelectrical Impedance Analysis. Weight and height will be combined to report BMI in kg/m^2
Change in lean mass | Baseline and 12 weeks
  Lean mass (kg) will be assessed using a dual-energy x-ray absorptiometer (DXA) and a TANITA's Bioelectrical Impedance Analysis.
Change in fat mass | Baseline and 12 weeks
  Fat mass (kg) will be assessed using a dual-energy x-ray absorptiometer (DXA) and a TANITA's Bioelectrical Impedance Analysis.
Change in bone mineral content and density | Baseline and 12 weeks
  Bone mineral content and density (z-score) will be assessed using a dual-energy x-ray absorptiometer (DXA).
Change in blood pressure | Baseline and 12 weeks
  Systolic and diastolic blood pressure will be assessed by a blood pressure monitor. Central blood pressure will be also analyzed using the SphygmoCor XCEL
Change in arterial stiffness | Baseline and 12 weeks
  Arterial stiffness will be assessed using the pulse wave analysis and pulse wave velocity determined by the SphygmoCor XCEL
Change in blood-based inflammatory biomarkers | Baseline and 12 weeks
  Blood samples will be used to determine plasmatic concentrations of inflammatory peripheral biomarkers including tumor necrosis factor-alpha (TNF-alpha) and interleukin-1 beta (IL-1beta), glucose, insulin, HDL and LDL cholesterol.
Change in saliva-based inflammatory biomarkers | Baseline and 12 weeks
  Saliva samples will be used to determine saliva concentrations of inflammatory peripheral biomarkers including tumor necrosis factor-alpha (TNF-alpha) and interleukin-1 beta (IL-1beta).
Change in blood-based cardiovascular biomarkers | Baseline and 12 weeks
  Blood samples will be used to determine plasmatic concentrations of cardiovascular peripheral biomarkers including glucose, insulin, HDL and LDL cholesterol.
Change in saliva-based cardiovascular biomarkers | Baseline and 12 weeks
  Saliva samples will be used to determine plasmatic concentrations of cardiovascular peripheral biomarkers including glucose, insulin, HDL and LDL cholesterol.
Change in epigenetics | Baseline and 12 weeks
  Blood samples will be stored for epigenetic analyses.
Change in gene expression | Baseline and 12 weeks
  Blood samples will be stored for genetic analyses, including APOE and BDNF genotypes.
Change in oral and gut microbiota | Baseline and 12 weeks
  Saliva and fecal samples will be used to determine oral and gut microbiota including the most representative phyla (i.e., firmicutes, bacteroidetes, and proteobacteria)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco B Ortega, Professor, Principal Investigator — Department of Physical Education and Sports, Faculty of Sport Sciences, University of Granada, Spain
Locations (1):
- Sport and Health University Research Institute (iMUDS), Technological Health Park, University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
The protocol, statistical analyses plan and data management plan will be share open access. Data files including IPD, and corresponding data dictionaries, will be shared under restricted access and upon reasonable request (contact FB Ortega) due to privacy issue and GDPR regulations. In principle, all collected IPD will be available for sharing under the "as open as possible, as closed as necessary" principle. The shared data files will be pseudonymized, only include participants who provided informed consent for sharing, and sharing is only possible when the data is used for research purposes regarding exercise, and cardiovascular and brain health. This is stated at the informed consent files that the participants signed when they agree to participate
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD data will be available 12 months after the primary outcome paper published. The data will be available 15 years after data collection.
Access Criteria: The specific process of data access will be determined in a later stage, but in general the research team supports data sharing. Roughly, data will be available upon reasonable request to the PI (FB Ortega). The data requests must contain the purpose and aim of the research, but also specification of the data requested, and data analysis before data sharing. Data will only be shared for research purposes on exercise, cardiovascular and brain health. In addition, we will follow "as open as possible, as closed as necessary" principle, so depending on this principle we will decide whether the data could be shared. A data access committee will be installed to approve data requests.

REFERENCES:
- [Background] Toval A, Solis-Urra P, Bakker EA, Sanchez-Aranda L, Fernandez-Ortega J, Prieto C, Alonso-Cuenca RM, Gonzalez-Garcia A, Martin-Fuentes I, Fernandez-Gamez B, Olvera-Rojas M, Coca-Pulido A, Bellon D, Sclafani A, Sanchez-Martinez J, Rivera-Lopez R, Herrera-Gomez N, Penafiel-Burkhardt R, Lopez-Espinosa V, Corpas-Perez S, Garcia-Ortega MB, Vega-Cordoba A, Barranco-Moreno EJ, Morales-Navarro FJ, Nieves R, Caro-Rus A, Amaro-Gahete FJ, Mora-Gonzalez J, Vidal-Almela S, Carlen A, Migueles JH, Erickson KI, Moreno-Escobar E, Garcia-Orta R, Esteban-Cornejo I, Ortega FB. Exercise and brain health in patients with coronary artery disease: study protocol for the HEART-BRAIN randomized controlled trial. Front Aging Neurosci. 2024 Aug 23;16:1437567. doi: 10.3389/fnagi.2024.1437567. eCollection 2024. PMID 39246594
- [Background] Toval A, Bakker EA, Granada-Maia JB, Nunez de Arenas-Arroyo S, Solis-Urra P, Eijsvogels TMH, Esteban-Cornejo I, Martinez-Vizcaino V, Ortega FB. Exercise type and settings, quality of life, and mental health in coronary artery disease: a network meta-analysis. Eur Heart J. 2025 Jun 16;46(23):2186-2201. doi: 10.1093/eurheartj/ehae870. PMID 39809303

DOCUMENTS (2):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT06214624/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT06214624/SAP_001.pdf